CLINICAL TRIAL: NCT02268500
Title: VAccination to Improve Clinical outComes in Heart Failure Trial (VACC-HeFT): a Feasibility Study
Brief Title: VAccination to Improve Clinical outComes in Heart Failure Trial: a Feasibility Study (VACC-HeFT)
Acronym: VACC-HeFT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2014-0656
Record Dates: First submitted 2014-10-08; First posted 2014-10-20 (Estimated); Results first posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Chronic Heart Failure
MeSH Terms: interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard dose influenza vaccine (Active Comparator): Standard dose (45ug) influenza vaccine will be administered intramuscularly
  Interventions: Biological: Influenza vaccine
- High dose influenza vaccine (Active Comparator): High dose (180ug) influenza vaccine will be administered intramuscularly
  Interventions: Biological: Influenza vaccine

INTERVENTIONS:
Biological: Influenza vaccine — Influenza vaccine
  Other Names: Fluzone

SUMMARY:
A multi-center, prospective, randomized, open-label blinded-endpoint trial in patients with heart failure will be conducted; 20 will be assigned to the standard dose vaccine dose and 20 patients to high dose influenza vaccine. Post-vaccine antibody measurements will be assessed, as well as tolerability differences between groups.

DETAILED DESCRIPTION:
This is a randomized, double blind, active-control trial of high dose influenza vaccine compared to standard dose influenza vaccine for one season in adult participants with symptomatic heart failure(HF). The primary outcome measure is humoral (antibody-mediated) immune response, and secondary outcomes include cumulative incidence of influenza-like illness symptoms and all cause hospitalizations. The aim is to gather information on feasibility of this study design and effect size differences to inform a larger outcomes-based clinical trial.

The 5.8 million Individuals in the US with heart HF are at high risk for influenza infection and associated morbidity, mortality and increased health care costs despite annual influenza vaccination. Higher dose of vaccine is approved for use in older adults. Antibody-mediated immunity contributes to vaccine-induced protection from influenza illness. Investigators at University of Wisconsin(UW) Madison have demonstrated reduced antibody titers to influenza vaccination in patients with HF. Additionally, study team has shown in a pilot study that double dose influenza vaccine resulted in increased titers and was well tolerated.

A multi-center, prospective, randomized, open-label blinded-endpoint trial will be conducted with 20 participants assigned to the standard dose vaccine dose and 20 participants to high dose influenza vaccine. The primary outcome measure is the rate of seroconversion (4-fold rise in antibody titers to A/H3N2, A/H1N1, and B-type vaccine antigens), assessed 4 weeks post vaccination. The study will also examine feasibility differences in symptoms of influenza and all-cause hospitalizations between vaccine dose groups, and these data will be used for planning a subsequent outcomes-based clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Adults > 18 years old
2. Able to give informed consent
3. Systolic or diastolic dysfunction
4. Previously or currently symptomatic heart failure
5. Stable on current heart failure drug therapy regimen for > 30 days and no change in heart failure drug therapy regimen on day of enrollment
6. Hospitalization (for any reason) in last 12 months
7. Received influenza vaccination the prior season

Exclusion Criteria:

1. History of allergic reaction or adverse event to influenza vaccine
2. Documented severe allergy to egg products
3. Unwilling or unable to give consent
4. Moderate to severe acute febrile illness at baseline
5. Immunologic conditions that may affect immune responses per clinical judgment of the investigators
6. Use of immunosuppressants or immunomodulating therapies within 3 months of the study, including prednisone, cyclosporine, tacrolimus, methotrexate, azathioprine, mycophenolate mofetil, cyclophosphamide, and injectable interferons
7. Participation in a clinical trial within 30 days
8. Absence for more than 7 consecutive days during the surveillance period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-09; Primary Completion 2016-01 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Orly Vardeny, PharmD, MS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Dose Influenza Vaccine | High Dose Influenza Vaccine
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Dose Influenza Vaccine | High Dose Influenza Vaccine | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (12.2) | 62.5 (13.1) | 59.45 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 17 | 21 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 23 | 24 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 24 | 23 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Left Ventricular Ejection Fraction (LVEF) percentage [Mean (Standard Deviation); unit: percentage of ejection fraction] | 38.8 (9.8) | 40.3 (10.2) | 39.55 (10)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 33.7 (10) | 30.9 (6.8) | 32.3 (8.4)
number of current tobacco users [Count of Participants; unit: Participants] | 1 | 1 | 2
Participants with Diabetes mellitus [Count of Participants; unit: Participants] | 4 | 11 | 15
Participants with Atrial fibrillation [Count of Participants; unit: Participants] | 12 | 9 | 21
Participants with Ischemic etiology [Count of Participants; unit: Participants] | 6 | 8 | 14
Aspirin users [Count of Participants; unit: Participants] | 12 | 20 | 32
Angiotensin converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB) users [Count of Participants; unit: Participants] | 23 | 23 | 46
Beta blocker users [Count of Participants; unit: Participants] | 22 | 23 | 45
Mineralocorticoid Receptor Antagonists (MRA) users [Count of Participants; unit: Participants] | 17 | 13 | 30
Diuretic users [Count of Participants; unit: Participants] | 20 | 19 | 39
Long acting nitrate users [Count of Participants; unit: Participants] | 1 | 1 | 2
Number of Digoxin users [Count of Participants; unit: Participants] | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 4 Fold Rise in Serum Antibody Concentration of A/H1N1 Vaccine Antigens
Time Frame: 4 weeks
Population: 1 participant from 'standard dose influenza vaccine' arm and 1 participant from 'high dose influenza vaccine' arm were excluded as the sample was inadequate to run the assay.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dose Influenza Vaccine | High Dose Influenza Vaccine
Number analyzed (Participants) | 23 | 23
Participants | 11 | 12
Statistical Analysis 1: Comparison: Standard Dose Influenza Vaccine vs High Dose Influenza Vaccine; Test type: Superiority; p = 0.89, Chi-squared

2. Primary Outcome: Number of Participants With 4 Fold Rise in Serum Antibody Concentration of A/H3N2 Vaccine Antigens
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dose Influenza Vaccine | High Dose Influenza Vaccine
Number analyzed (Participants) | 23 | 23
Participants | 15 | 17
Statistical Analysis 1: Comparison: Standard Dose Influenza Vaccine vs High Dose Influenza Vaccine; Test type: Superiority; p = 0.43, Chi-squared

3. Primary Outcome: Number of Participants With 4 Fold Rise in Serum Antibody Concentration of B-type Vaccine Antigens
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dose Influenza Vaccine | High Dose Influenza Vaccine
Number analyzed (Participants) | 23 | 23
Participants | 7 | 14
Statistical Analysis 1: Comparison: Standard Dose Influenza Vaccine vs High Dose Influenza Vaccine; Test type: Superiority; p = 0.03, Chi-squared

4. Secondary Outcome: Number of Participants With Influenza Like Illness
Description: Influenza Like Illness is not considered adverse event.
Time Frame: 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dose Influenza Vaccine | High Dose Influenza Vaccine
Number analyzed (Participants) | 24 | 24
Participants | 8 | 7
Statistical Analysis 1: Comparison: Standard Dose Influenza Vaccine vs High Dose Influenza Vaccine; Test type: Superiority; p = 0.76, Chi-squared

5. Secondary Outcome: Number of All-cause Hospitalizations
Description: All-cause hospitalizations are not considered adverse events.
Time Frame: 8 months
Measure: Number; unit: hospitalizations
Arm/Group | Standard Dose Influenza Vaccine | High Dose Influenza Vaccine
Number analyzed (Participants) | 24 | 24
hospitalizations | 15 | 6
Statistical Analysis 1: Comparison: Standard Dose Influenza Vaccine vs High Dose Influenza Vaccine; Test type: Superiority; p = 0.01, Chi-squared

ADVERSE EVENTS:
Time Frame: 1 week
Description: 1 week post randomization, participants were contacted by phone for ascertainment of injection related adverse events.
Arm/Group | Standard Dose Influenza Vaccine | High Dose Influenza Vaccine
All-Cause Mortality (participants affected / at risk) | 1/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes